CLINICAL TRIAL: NCT02494869
Title: Dose-Response of Aerobic Training in Women at High-Risk for Development of Breast Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15-093
Record Dates: First submitted 2015-07-08; First posted 2015-07-10 (Estimated); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: High Risk for Developing Breast Cancer
Keywords: Aerobic Training; Exercise; Gene Expression; 15-093
MeSH Terms: conditions — Motor Activity | interventions — Body Height; Weights and Measures; Blood Specimen Collection; Exercise Test

ARMS (4):
- Nonlinear Aerobic Training (75 minutes/week) closed to accrual (Experimental): The ultimate goal is for participants to complete 75 minutes/week of structured aerobic training per week at 55% to 100% of the individually determined exercise capacity (VO2peak) determined from the (CPETs performed at baseline, midpoint, and Study Follow-Up. The 75 min/wk will be achieved via 3 individual supervised aerobic training sessions at approximately 25 minutes/session.All other on- site participants in Arms A and B will be provided with a heart rate monitor to thank them for completing the study. This arm is closed to accrual.
  Interventions: Behavioral: Nonlinear Aerobic Training; Other: Height, Weight, BMI measure; Other: Blood draw; Other: Cardiopulmonary exercise test
- Nonlinear Aerobic Training (150 minutes/week) (Experimental): The ultimate goal is for participants to complete 150 minutes/week of structured aerobic training per week at 55% to 100% of the individually determined exercise capacity (VO2peak) determined from the CTPETs test performed at baseline, midpoint, and Study Follow-Up. The 150 minutes/week will be achieved by completing 3 aerobic training sessions/week for approximately 50 minutes/session. All other on- site participants in Arms A and B will be provided with a heart rate monitor to thank them for completing the study.
  Interventions: Behavioral: Nonlinear Aerobic Training; Other: Height, Weight, BMI measure; Other: Blood draw; Other: Cardiopulmonary exercise test
- Nonlinear Aerobic Training (300 minutes/week) (Experimental): The ultimate goal is for participants to complete 300 minutes/week of aerobic training per week at 55% to 100% of the individually determined exercise capacity (VO2peak) determined from CPETs performed at baseline, midpoint, and Study Follow-Up. The 300 minutes/week will be achieved by completing 5 aerobic training sessions/week for approximately 60 minutes/session. A minimum of 3 sessions/week are required to be supervised while the remaining 2 sessions can be supervised or unsupervised home-based. Participants on all Arms will receive a heart rate monitor prior to beginning unsupervised home-based aerobic training sessions. Vital sign monitoring guidelines for unsupervised sessions, prescribed at lower intensities, will be advised by the exercise physiologist at the time the session plan is provided to the patient. Patients will be instructed to not begin an unsupervised session if their resting heart rate or blood pressure is outside the recommended guidelines.
  Interventions: Behavioral: Nonlinear Aerobic Training; Other: Height, Weight, BMI measure; Other: Blood draw; Other: Cardiopulmonary exercise test
- General Physical Activity (Active Comparator): Usual care patients will receive a home-based, general physical activity program. Specifically, all patients assigned to general physical activity will receive an initial, in-person consultation with staff exercise physiologist outlining a structured home-based aerobic walking program with a goal up to 150 minutes per week outside of their normal daily activity. Patients can be provided with a fitness tracker (e.g. FitBit) to evaluate exercise duration and intensity. Patients may also be provided with an exercise log to records type, duration, and average heart rate during sessions. The exercise log is provided as a guidance tool and may be, although is not required to be, returned to study staff. Staff exercise physiologists will contact patients to check progress and answer questions.
  Interventions: Other: Blood draw

INTERVENTIONS:
Behavioral: Nonlinear Aerobic Training
  Arms: Nonlinear Aerobic Training (150 minutes/week); Nonlinear Aerobic Training (300 minutes/week); Nonlinear Aerobic Training (75 minutes/week) closed to accrual
Other: Height, Weight, BMI measure
  Arms: Nonlinear Aerobic Training (150 minutes/week); Nonlinear Aerobic Training (300 minutes/week); Nonlinear Aerobic Training (75 minutes/week) closed to accrual
Other: Blood draw
Other: Cardiopulmonary exercise test
  Arms: Nonlinear Aerobic Training (150 minutes/week); Nonlinear Aerobic Training (300 minutes/week); Nonlinear Aerobic Training (75 minutes/week) closed to accrual

SUMMARY:
This study is being done to look at the effect that different amounts of progressive exercise training has on risk factors associated with developing breast cancer. These risk factors include exercise capacity, body weight, and body composition, as well as the expression of certain genes and levels of inflammatory factors in your breast tissue.

The participant will be instructed to self-report the session information to ExOnc staff at or before their next scheduled visit. If the participant's next scheduled visit is greater than 72 hours following an unsupervised session, ExOnc staff may reach out to the participant to retrieve the session information. Unsupervised session details will be source documented by ExOnc staff.

ELIGIBILITY:
Inclusion Criteria:

* Women at high-risk of breast cancer as defined by one of the following:

  * Cytologically confirmed atypical hyperplasia
  * Cytologically confirmed LCIS
* Being a carrier for

  * BRCA1 and/or BRCA2
  * Predicted lifetime risk of breast cancer >20% based on family history)
  * Predicted 10-year risk of breast cancer of ≥ 2.31%
  * Predicted 5-year risk of breast cancer ≥ 1.67%
  * Aged 21 ≤ 80 years old
  * If a female of child-bearing potential, must not be pregnant or planning to become pregnant during the study.
  * Women <50 years old who are of child-bearing potential must have a negative pregnancy test (urine HCG or serum) within 14 days of enrollment.
* Must a negative mammogram or negative breast MRI within 1 year of protocol required baseline core biopsy
* Clinical breast exam interpreted as benign (not suspicious for cancer) at MSK
* Performing less than or equal to 120 minutes of structured moderate-intensity or strenuous-intensity exercise per week
* Able to complete an acceptable baseline CPET in the absence of high risk ECG findings or other inappropriate response to exercise as determined by the investigator.
* Able to achieve an acceptable peek baseline CPET defined as by any of the following criteria:

  * achieving a plateau in oxygen consumption concurrent an with increase in power output;
  * a respiratory exchange ratio ≥ 1.10;
  * attainment of maximal predicted heart rate (HRmax) (i.e., within 10 bpm of age-predicted [HRmax = 220-Age[years]) Volitional exhaustion, as measured by a rating of perceived exertion (RPE) ≥ 18 on the BORG scale.

Exclusion Criteria:

* Use of any selective estrogen receptor modulator or aromatase inhibitor within 6 months of randomization, including, but not limited to: (tamoxifen, raloxifene, arzoxifene, acolbifene, anastrozole, exemestane, and letrozole)
* Enrollment on an interventional investigational study
* Bilateral breast implants
* Any newly identified breast abnormality requiring surgical excision
* History of any of the following:
* Invasive cancer diagnosis
* DCIS
* Any current invasive cancer diagnosis
* Metastatic malignancy of any kind
* Any other condition or intercurrent illness that in the opinion of the investigator makes the subject a poor candidate for core biopsy or the trial
* Mental impairment leading to inability to cooperate.
* Room air desaturation at rest ≤85%
* Any of the following absolute contraindications to cardiopulmonary exercise testing and/or aerobic training:
* Acute myocardial Infarction (within 3-5 days of any planned study procedures);
* Unstable angina;
* Uncontrolled arrhythmia causing symptoms or hemodynamic compromise;
* Recurrent syncope;
* Active endocarditis;
* Acute myocarditis or pericarditis;
* Symptomatic severe aortic stenosis;
* Uncontrolled heart failure;
* Acute pulmonary embolus or pulmonary infarction within 3 months of any planned study procedures;
* Thrombosis of lower extremities;
* Suspected dissecting aneurysm;
* Uncontrolled asthma;
* Pulmonary edema;
* Respiratory failure;
* Acute non-cardiopulmonary disorders that may affect exercise performance or be aggravated by exercise (i.e. infection, renal failure, thyrotoxicosis); or

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women at High-Risk for Development of Breast Cancer
Enrollment: 75 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
gene expression patterns of non-neoplastic breast epithelial cells in women at high-risk for development of breast cancer | 2 years
  Fresh-frozen tissue sections from normal breast epithelial cell samples before and after aerobic training will be cut and stained using hematoxylin & eosin, and the morphological features will be reviewed.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Scott, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/